CLINICAL TRIAL: NCT05429463
Title: Neoadjuvant Therapy of Sintilimab Combined With Chemotherapy for Resectable Squamous Cell NSCLC（neoSCORE Ⅱ）：A Prospective, Randomized, Open-Label, Multi-Center Phase 3 Trial
Brief Title: Neoadjuvant Therapy of Sintilimab Combined With Chemotherapy for Resectable Squamous Cell NSCLC（neoSCORE Ⅱ）
Acronym: neoSCORE Ⅱ
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: neoSCORE Ⅱ
Record Dates: First submitted 2022-06-19; First posted 2022-06-23 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Squamous Cell Non-small Cell Lung Cancer
Keywords: Sintilimab; Squamous Cell NSCLC; Neoadjuvant immunochemotherapy
MeSH Terms: interventions — sintilimab; spartalizumab; Carboplatin; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A(3 cycles of neoadjuvant therapy) (Experimental): Neoadjuvant: Prior to surgery, participants receive up to 3 cycles (cycle length: 3 weeks) of sintilimab [200 mg, intravenous (IV); given on cycle day 1] in combination with neoadjuvant chemotherapy, consisting of albumin-bound paclitaxel [260 mg/m^2, IV; given on cycle day 1] and carboplatin [AUC 5- 6mg/mL/min, IV; given on cycle day 1 ] .
  Adjuvant: Followed by surgery within the 3-5th week after the last dose of sintilimab, the researcher will decide whether to radiotherapy or not according to the clinical situation and pathological stage of the patient. The maintenance treatment of sintilimab [200 mg, intravenous (IV); given on cycle day 1; cycle length: 3 weeks] may be selected upon subject request for up to 1 year.
  Interventions: Biological: Sintilimab; Drug: Carboplatin; Drug: Albumin-Bound Paclitaxel
- Arm B(4 cycles of neoadjuvant therapy) (Experimental): Neoadjuvant: Prior to surgery, participants receive up to 4 cycles (cycle length: 3 weeks) of sintilimab [200 mg, intravenous (IV); given on cycle day 1] in combination with neoadjuvant chemotherapy, consisting of albumin-bound paclitaxel [260 mg/m^2, IV; given on cycle day 1] and carboplatin [AUC 5- 6mg/mL/min, IV; given on cycle day 1 ] .
  Adjuvant: Followed by surgery within the 3-5th week after the last dose of sintilimab, the researcher will decide whether to radiotherapy or not according to the clinical situation and pathological stage of the patient. The maintenance treatment of sintilimab [200 mg, intravenous (IV); given on cycle day 1; cycle length: 3 weeks] may be selected upon subject request for up to 1 year.
  Interventions: Biological: Sintilimab; Drug: Carboplatin; Drug: Albumin-Bound Paclitaxel

INTERVENTIONS:
Biological: Sintilimab — 200 mg by IV infusion every 3 weeks (Q3W), given on cycle day 1.
  Other Names: IBI308; PD-1 antibody
Drug: Carboplatin — AUC 5-6 mg/mL/min by IV infusion Q3W, given on cycle day 1.
Drug: Albumin-Bound Paclitaxel — 260 mg/m^2 by IV infusion Q3W, given on cycle day 1.

SUMMARY:
This is a Phase 3, prospective, randomized, open-label, multi-center study that assesses the efficacy and safety of neoadjuvant therapy with different cycles of sintilimab combined with chemotherapy for Resectable Squamous Cell NSCLC. This trial will also explore the biomarkers of neoadjuvant immunochemotherapy.

DETAILED DESCRIPTION:
This is a Phase 3, prospective, randomized, open-label, multi-center study that assesses the efficacy and safety of neoadjuvant therapy with different cycles of sintilimab combined with chemotherapy for Resectable Squamous Cell NSCLC. In this trial, eligible subjects will be randomly assigned to arm A and arm B (1:1). Subjects in arm A will receive 3 cycles of neoadjuvant sintilimab with chemotherapy and arm B will receive 4 cycles of neoadjuvant sintilimab with chemotherapy, followed by surgery within the 3-5th week after the last dose of sintilimab. After operation, both subjects in arm A and B can receive the treatment of sintilimab for up to 1 year according to the requirements of patients. The primary purpose is MPR rate of Resectable Squamous Cell NSCLC with different cycles of sintilimab combined with chemotherapy, which is defined as the percentage of participants having ≤10% viable tumor cells in the pathological examination of resected specimens.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before starting any trial related procedure.Be willingness and able to undergo planned visits, protocol therapy, laboratory tests and other testing procedures.
2. 18-75 years old, male or female.
3. Squamous Cell Non-small cell lung cancer confirmed by cytology or histology.
4. There must be at least one evaluable focus judged according to recist1.1 standard.
5. Evaluation by the researchers and classified by the 8th version of AJCC TNM staging to confirm resectable stage cⅡA-ⅢB squamous NSCLC patients without any treatment before.
6. ECOG PS 0-1.
7. Life expectancy > 6 months.
8. Adequate organ function and it should meet the following criteria:

   Absolute value of neutrophils (ANC) ≥1.5×109/L in the absence of granulocyte colony stimulating factor for the past 14 days; Platelet ≥100×109/L in the last 14 days without blood transfusion; Hemoglobin >9g/dL in the absence of blood transfusion or erythropoietin in the last 14 days ;

   Total bilirubin(TBIL)≤1.5ULN, ALT、AST≤ 2.5 ULN, serum creatinine(sCr)≤1.5ULN;

   Good blood coagulation: INR≤1.5 or PT≤1.5 ULN;

   Normal thyroid function: TSH within normal institutional limits;
9. For women of reproductive age, a urine or serum pregnancy test with negative results should be performed within 3 days prior to receiving the first study drug administration (day 1 of cycle 1). If a urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is requested. Women of nonreproductive age were defined as at least 1 year after menopause or having undergone surgical sterilization or hysterectomy. If there is a risk of conception, all subjects (both men and women) will use a medically approved highly effective contraceptive (e.g., an intrauterine device, birth control pill, or condom) for the entire treatment period up to 120 days after the last study drug (or 180 days after the last chemotherapy drug).

Exclusion Criteria:

1. Malignancies within 5 years prior to the first dose(excluding radical skin basal cell carcinoma, skin squamous cell carcinoma and / or radical resection of carcinoma in situ).
2. Currently participating in the intervention clinical treatment, or receiving other drugs or research instruments within 4 weeks before the first dose.
3. Patients who have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or drugs for another stimulation or synergistic inhibition of T cell receptor (e.g. CTLA-4, OX-40, CD137).
4. Active autoimmune diseases requiring systemic treatment (e.g. using disease improving drugs, corticosteroids or immunosuppressants) occurred within 2 years before the first dose. Alternative therapies (e.g. thyroxine, insulin or corticosteroids in physiological doses for adrenal or pituitary insufficiency) are not considered systemic treatment.
5. Systemic glucocorticoid therapy (excluding local glucocorticoids by nasal spray, inhalation or other routes) or any other form of immunosuppressive therapy is in progress within 7 days before the first dose.

   Note: it is allowed to use physiological dose of glucocorticoid (Prednisone≤10 mg/d or equivalent drug).
6. Received allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
7. Allergic to study drug(sintilimab, carboplatin, albumin-bound paclitaxel) components excipients.
8. Not fully recovered from toxicity and/ or complications caused by any intervention before treatment (≤level 1 or reach baseline, excluding fatigue or hair loss).
9. Has a known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibody positive).
10. Untreated active Hepatitis B (defined as HBsAg positive and HBV-DNA copies>ULN).
11. Active Hepatitis C (HCV antibody positive and HCV-RNA level higher than the detection limit).
12. Inoculate the live vaccine within 30 days before the first dose (cycle 1 day 1).

    Note: it is allowed to receive the injection inactivated virus vaccine for seasonal influenza within 30 days before the first dose; however, it is not allowed to accept the live attenuated influenza vaccine for intranasal medication.
13. Pregnant or lactating women.
14. There are any serious or uncontrollable systemic diseases, such as:

    Resting ECG has significant abnormalities in rhythm, conduction or morphology, and the symptoms are serious and difficult to control,such as complete left bundle branch block, heart block above degree Ⅱ, ventricular arrhythmia or atrial fibrillation;

    Unstable angina, congestive heart failure, chronic heart failure with NYHA grade ≥ 2;

    Within 6 months before inclusion, there were any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic attack etc;

    History of noninfectious pneumonia requiring glucocorticoid treatment within 1 year before the first dose,or having currently clinical active interstitial lung diseases;

    Active pulmonary tuberculosis;

    Active or uncontrolled infections requiring systemic treatment;

    Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;

    Poorly controlled diabetes (Fasting blood glucose (FBG)>10mmol/L);

    Urine routine test indicates that urine protein≥++, and confirmed that 24 hours proteinuria>1.0 g;

    Patients with mental disorders who are unable to cooperate with the treatment;
15. There are medical history, disease, treatment or laboratory abnormal results that may interfere with the test results, prevent the subjects from participating in the whole process of the study, or the researchers think that participating in the study is not in the best interests of the subjects or there are other potential risks that the subjects are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-11-11 (Estimated); Study Completion 2029-11-11 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate (MPR) | At time of surgery
  MPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the pathological examination of resected specimens.

SECONDARY OUTCOMES:
Pathology complete response rate(pCR) | At time of surgery
  pCR rate is defined as the percentage of participants lacking of evidence of viable tumor cells in the pathological examination of resected specimens.
Objective response rate (ORR) | prior to surgery
  ORR is defined as the percentage of participants having a complete response or a partial response, measured by RECIST 1.1.
2 years disease-free survival rate (DFS) | 2 years postoperatively
  2 years DFS rate is defined as the percentage of participants having no recurrence, distant metastasis or death within 2 years after operation.
2 years overall survival rate (OS) | 2 years postoperatively
  2 years OS rate is defined as the percentage of participants having no death of any cause within 2 years after operation.The Kaplan-Meier estimator will be used to estimate median OS and its 95%CI and the survival curve.
2 years event free survival (EFS) | 2 years after randomization
  2 years EFS rate is defined as the percentage of participants having no radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause within 2 years after randomization.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Shao M, Yao J, Zhao L, Li L, Chen M, Zhang Y, Liu H, Chen Z, Li B, Wu Z, Fan J, Qiu F. NeoSCORE II: three vs four cycles of neoadjuvant sintilimab + chemotherapy for squamous non-small-cell lung cancer. Future Oncol. 2024 Jan;20(3):121-129. doi: 10.2217/fon-2024-0026. Epub 2024 Feb 14. PMID 38353107